CLINICAL TRIAL: NCT00838760
Title: Phase I, Double-blind, Randomized, Placebo-controlled Trial to Examine the Safety, Tolerability and Plasma Pharmacokinetics of Increasing Single Oral Doses of TMC558445 With and Without Food, and Increasing Repeated Oral Doses in Combination With a Single Dose of TMC310911
Brief Title: PEPI-TiDP23-C103: First-in-Human Study to Examine the Safety, Tolerability, and Plasma Pharmacokinetics of Increasing Single and Repeated Oral Doses of TMC558445 and of a Combined Single Day Dosing of Oral TMC558445 and Oral TMC310911 and Also Oral Darunavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Compound Development Team Leader, Tibotec Pharmaceuticals, Ireland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR015955
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: HIV-1
Keywords: PEPI-TiDP23-C103; PEPI-C103; PEPI; TMC558445; TMC310911; Darunavir, Healthy volunteers; Pharmacokinetics; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — TMC-310911; Darunavir

INTERVENTIONS:
Drug: TMC558445; TMC310911; Darunavir; Placebo

SUMMARY:
The purpose of the study is to determine the safety, tolerability and plasma pharmacokinetics (pk) (i.e., the levels of TMC558445 circulating in your blood over time) of increasing single oral doses of TMC558445 and of multiple increasing oral doses followed by a single dose of TMC310911 to assess the potential boosting effect on the latter compound. In this study, two investigational new drugs are involved, TMC558445 and TMC310911.

The study has been amended as follows:

TMC558445 will be administered either twice a day (b.i.d.) or once daily (q.d.). A single 300 mg or 600 mg dose of TMC310911 will be administered under fasted or fed conditions. The boosting effect on Darunavir will be investigated.

DETAILED DESCRIPTION:
This is a First-in-Human Phase I, double-blind (neither physician or patient knows the name of the assigned study drug), randomized (study medication assigned by chance), placebo-controlled trial for TMC558445 to examine the safety, tolerability and plasma pharmacokinetics after increasing single oral doses of TMC558445 and after increasing oral repeated doses of TMC558445, followed by a single day dosing of TMC558445 and TMC310911. This combination will assess the potential pharmacokinetic enhancement (boosting) on the latter compound. TMC558445 is to be used as a booster for TMC310911. The trial consists of 2 parts: a single dose escalation and a multiple dose escalation part. The single dose escalation part will consist of 6 sessions. The single dose part will include 18 healthy adult volunteers, divided over 2 panels. In each session, 6 healthy volunteers will receive TMC558445 and 3 healthy volunteers will receive placebo with standard meals. Intake of TMC558445/placebo will take place on Day 1 of each session between 07:00 and 11:00 a.m. Single doses of 40, 100, 200, 400, 800, and 1600 mg of TMC558445/placebo will be administered alternating over the 2 panels. The trial will be stopped earlier when the maximum tolerated dose is reached. A washout period (a period where no treatment will be taken in view of having all the medication eliminated from the body before starting a new treatment) of at least 10 days will be respected between consecutive TMC558445/placebo dosings. Once, a food effect will be studied under fasted conditions at one of the previously studied doses. The multiple dose escalation part of this trial will start when the 200 mg dose is found to be safe.This part of the trial will include 27 healthy adult volunteers, divided over 3 panels: 6 will receive TMC558445 and 3 will receive placebo. TMC558445/placebo will be administered during 7 consecutive days. The treatment will be twice daily between 07:00 and 11:00 a.m. and between 07:00 and 11:00 p.m. Volunteers will receive a single oral dose of 300 mg of TMC310911 on Day 7 and on Day 1 of Session XI (after a washout period of at least 14 days). Dose escalation in the single and multiple ascending dose regimens will continue only if the previous dose was found safe. Pharmacokinetic profiles of TMC558445 will be determined up to a max of 72 h after the last intake per session. Pharmacokinetic profiles of TMC310911 will be determined over 24 h. The expected duration of the investigational period in the single escalation dose part is at least 8 weeks and at least 3 weeks in the multiple escalation dose part. Safety and tolerability evaluations will be recorded at regular intervals throughout the trial. Blood and urine samples will be taken at predefined timings as well as ECG measurements, vital signs (blood pressure and heart rate), and physical examinations. The study has been amended. In Panel 5, TMC558445 may now be administered either twice daily or once daily and TMC310911 may be given at a 300 mg or 600 mg single dose. Decision on dosing regimen, TMC310911 dose and food conditions will be made based on results of the previous panels.

The study has been amended as follows:

Panel 6 (9 adult volunteers), will receive 800 mg Darunavir (DRV) on day 7 combined with TMC55844 that has been given for 7 days at 200 mg once daily dosis. After a wash out period of 14 days the participants will receive Darunavir 800 mg alone. TMC558445, TMC310911 or placebo will be formulated as oral drinkable solution. Part 1 will consist of single dose TMC558445/placebo from 40 up to 1600mg on Day 1 of each session with a volume between 2 and 20ml. Part 2 will consist of TMC558445/placebo twice daily from Day 1 to Day 7 with max dose of 200mg and volume of 5 ml + a single intake of 300 or 600mg TMC310911(12/24ml)/ DRV 800mg on morning of Day 7 in one session and single dose of TMC310911/ DRV on Day 1 in the second session.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmokers for at least 3 months prior to selection
* Weight as defined by a Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included
* Informed Consent Form (ICF) signed voluntarily
* Able to comply with protocol requirements
* Healthy on the basis of a pretrial physical examination, medical history, the results of blood biochemistry and hematology tests, a urinalysis, vital signs, and a 12-lead electrocardiogram (ECG)

Exclusion Criteria:

* Past history of clinically significant heart arrhythmias (extrasystoli, tachycardia at rest)
* Having baseline prolongation of QTc interval > 450 ms, history of risk factors for Torsade de Pointes syndrome (hypokalemia, family history of long QT Syndrome)
* Female, except if postmenopausal for more than 2 years, or post-hysterectomy or post-surgical sterilization (without reversal operation)
* Currently active clinically relevant or significant underlying gastrointestinal, cardiovascular, nervous system, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease
* History of clinically relevant skin disease or allergy including drug allergy as well

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The trial objectives are to determine the safety, tolerability and plasma pharmacokinetics of TMC558445 after increasing single oral doses from 40 mg up to 1600 mg or up to the MTD and after increasing multiple oral doses at 3 dose levels. | safety & tolerability will be determined throughout the study. PK profiles of TMC558445 will be determined up to a max of 72 h after the last intake per session. Pk profiles of TMC310911/ DRV will be determined over 24 h.

SECONDARY OUTCOMES:
To determine the potential food effect on a single oral dose of TMC558445 at one dose level | 4 days
The safety and tolerability and the plasma pharmacokinetics of the repeated dosing for 7days of TMC558445 and a single 300 or 600mg dose of TMC310911 on Day7 | 7 days
The safety and tolerability and the plasma pharmacokinetics of the repeated dosing for 7days of TMC558445 and a single 800mg dose of DRV on Day7 | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited